CLINICAL TRIAL: NCT02861742
Title: Evaluation of the Impact of Emotional Skills of Young Women (≤ 45 Years), With Non-metastatic Breast Cancer, and Their Partner on Adjustment to Cancer
Brief Title: Impact of Emotional Skills of Young Women and Their Partner on Adjustment to Cancer
Acronym: KALICOU3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Université Lille 3 (Unknown); Aix Marseille Université (Other); University of Paris 5 - Rene Descartes (Other); SIRIC ONCOLille (Unknown); Canceropôle Nord Ouest (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KALICOU 3-1509; 2015-A01808-41 (Other: ANSM)
Record Dates: First submitted 2016-07-29; First posted 2016-08-10 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Aging; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study procedure (Other): Delivery of questionnaires, Questionnaire T1 to fill, Questionnaire T2 to fill, Questionnaire T3 to fill, Questionnaire T4 to fill, Questionnaire T5 to fill
  Interventions: Other: Delivery of questionnaires; Behavioral: Questionnaire T1 to fill; Behavioral: Questionnaire T2 to fill; Behavioral: Questionnaire T3 to fill; Behavioral: Questionnaire T4 to fill; Behavioral: Questionnaire T5 to fill

INTERVENTIONS:
Other: Delivery of questionnaires — After patient and partner information, clinical research associate or clinical research nurse will give to the couple 2 booklets containing 5 questionnaires, respectively T1, T2, T3, T4 and T5.
Behavioral: Questionnaire T1 to fill — T1 is to fill before chemotherapy.
Behavioral: Questionnaire T2 to fill — T2 is to fill after the 6th cycle of chemotherapy.
Behavioral: Questionnaire T3 to fill — T3 is to fill at the end of radiotherapy.
Behavioral: Questionnaire T4 to fill — T4 is to fill 4 month after beginning of hormonotherapy or surveillance if no hormonotherapy.
Behavioral: Questionnaire T5 to fill — T5 is to fill 1 year after the beginning of hormonotherapy or surveillance if no hormonotherapy.

SUMMARY:
The KALICOU 3 study will evaluate the effect of emotional skills of patients and their partners on their individual disease subjective experience during care pathways, from chemotherapy to surveillance.

DETAILED DESCRIPTION:
All women with breast cancer have to face, at any age, to numerous issues linked to cancer (incertitude, recurrence anxiety...) and to physical and psychosocial side effects of treatments which can degrade their life quality. However, young women (<45 years at diagnostic) have to face specific issues related to their age (early menopause, withdrawal of pregnancy projects, education of young children). Moreover, treatment consequences can alter patient's life quality and can persist in time (fatigue, pains, chemotherapy, sexuality, induced menopause for example). Overall, young patients have a lesser life quality, greater emotional distress and vulnerability and have more difficulties to establish adapted adjustment strategy compared to elder women.

The role and importance of relatives, particularly partners, during cancer pathology is incontestable. However, few empiric and consensual data exist on the impact of cancer diagnostic on partners, especially when women are young at initial diagnostic. Nevertheless, available data underline the importance of the supporting partner during breast cancer disease.

Cancer also disturbs conjugal relationship. For example, life quality of patient influence strongly the life quality and mental well-being of her partner. Moreover, the intimate relation with the partner could play an important role in healing after breast cancer. Numerous authors underline the importance of focus on the couple instead of patients alone or partners alone with a dyadic approach where dyad member's reactions will be interdependent.

Thus, study of dyadic adjustment of couples where a member is facing cancer pathology at young age is indubitably innovative and present a real scientific and clinical interest. More precisely, KALICOU 3 study will focus on the impact of intrapersonal and interpersonal emotional skills of patients and partners on individual and dyadic adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Patient and partner ≥ 18 years.
* Patient ≤ 45 years at diagnostic of non metastatic breast cancer.
* Disease relevant for neoadjuvant or adjuvant chemotherapy following or not by radiotherapy or hormonotherapy.
* Heterosexual or homosexual couples in a relationship since at least 6 months at the date of inclusion
* Patient affiliate to french social welfare system
* Informed consent sign by patient and partner before any study procedure

Exclusion Criteria:

* Psychological or physical inability to fill questionnaire
* Patient under guardianship

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2016-07-25 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
BCI-YW ( Breast Cancer Inventory - Young Women) | an average of 1 year
  To evaluate the effect of emotional skills of patients and partners on their individual disease subjective experience during care pathways, from chemotherapy to surveillance
BCI-Partner's YW ( Breast Cancer Inventory - Young Women Partner's) | an average of 1 year
  To evaluate the effect of emotional skills of patients and partners on their individual disease subjective experience during care pathways, from chemotherapy to surveillance
PEC (Profile of Emotional Competences) | an average of 1 year
  To evaluate the effect of emotional skills of patients and partners on their individual disease subjective experience during care pathways, from chemotherapy to surveillance

SECONDARY OUTCOMES:
BCI-YW | an average of 1 year
  To evaluate the dyadic effect's emotional skills and treatment repercussion on adjustment to cancer as well as on partner
BCI-Partner's YW | an average of 1 year
  To evaluate the dyadic effect's emotional skills and treatment repercussion on adjustment to cancer as well as on partner
SF 36 (Short Form 36 - Health Survey) | an average of 1 year
  To evaluate the dyadic effect's emotional skills and treatment repercussion on adjustment to cancer as well as on partner
Hospital Anxiety-Depression Scale | an average of 1 year
  To evaluate the dyadic effect's emotional skills and treatment repercussion on adjustment to cancer as well as on partner
Profile of Emotional Competences | an average of 1 year
  To evaluate the dyadic effect's emotional skills on adjustment to cancer as well as on partner
MAVA (Measure of affectivity: Valence/Activation) | an average of 1 year
  To evaluate the dyadic effect's emotional skills on adjustment to cancer as well as on partner

CONTACTS AND LOCATIONS:
Overall Officials: VANLEMMENS Laurence, MD, Principal Investigator — Oscar Lambret; Christophe Véronique, Pr, Study Director — Université Lille 3
Locations (33):
- France (33):
  - ICO-Site Paul Papin, Angers
  - Centre Marie Curie, Arras
  - Institut Sainte Catherine, Avignon
  - Centre Pierre Curie - SCP de radiologie et d'imagerie médicale, Beuvry
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH de BOULOGNE-SUR-MER, Boulogne-sur-Mer
  - Centre François Baclesse, Caen
  - Centre Hôpitalier de Compiègne Noyon, Compiègne
  - Centre Léonard de Vinci, Dechy
  - Centre Georges François Leclerc, Dijon
  - CHU de Grenoble, Grenoble
  - Centre Hospitalier André Mignot, Le Chesnay
  - Centre Bourgogne, Lille
  - Centre Oscar Lambret, Lille
  - CHRU de Lille, Lille
  - Institut Paoli Calmettes, Marseille
  - Centre Gray, Maubeuge
  - ICM Val d'Aurelle, Montpellier
  - Le Confluent - Centre Catherine de Sienne, Nantes
  - CHU, Poitiers
  - CH René Dubos, Pontoise
  - ICC Reims, Reims
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Hôpital Privé des Côtes d'Armor, Saint-Brieuc
  - Institut curie-Hôpital Huguenin, Saint-Cloud
  - ICO- Istitut Gauducheau, Saint-Herblain
  - Unité d'Oncologie et d'hématologie ONCOSUD, Toulouse
  - CHU Bretonneau, Tours
  - Centre de Cancérologie des Dentellières, Valenciennes
  - CH Valenciennes, Valenciennes
  - Hôpital Privé de Villeneuve d'Ascq, Villeneuve-d'Ascq

IPD SHARING:
Plan to Share IPD: No